CLINICAL TRIAL: NCT02879955
Title: Effects of Carbohydrates on Gut Hormone Secretion After Gastric Bypass Surgery
Brief Title: Carbohydrates and Gut Hormones After Gastric Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Christoffer Martinussen, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CM-CARB-16
Record Dates: First submitted 2016-08-11; First posted 2016-08-26 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Overweight
Keywords: Glucagon-Like Peptide 1; Carbohydrates; Gastric bypass; Bariatric Surgery; Overweight
MeSH Terms: conditions — Overweight | interventions — Glucose; Fructose; Sucrose; isomaltulose; Acarbose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 gastric bypass operated patients (Experimental): 4 different carbohydrate loads ingested at separate study days will be tested against each others ability to induce GLP-1 secretion.
  Interventions: Other: Glucose + Fructose; Other: Sucrose; Other: Isomaltulose; Other: Sucrose + Acarbose
- 10 healthy control subjects (Experimental): 4 different carbohydrate loads ingested at separate study days will be tested against each others ability to induce GLP-1 secretion.
  Interventions: Other: Glucose + Fructose; Other: Sucrose; Other: Isomaltulose; Other: Sucrose + Acarbose

INTERVENTIONS:
Other: Glucose + Fructose — Ingestion of the separate monosaccharides glucose (25 g) and fructose (25 g) dissolved in 200 mL of water. The load provides 0.1385 mol glucose and 0.1385 mol fructose.
Other: Sucrose — Ingestion of the disaccharide sucrose (47.5 g) dissolved in 200 mL of water. The load provides 0.1385 mol glucose and 0.1385 mol fructose.
Other: Isomaltulose — Ingestion of the slowly digestable disaccharide isomaltulose (47.5 g) dissolved in 200 mL of water. The load provides 0.1385 mol glucose and 0.1385 mol fructose.
Other: Sucrose + Acarbose — Ingestion of the disaccharide sucrose (47.5 g) and the alpha glucosidase inhibitor acarbose dissolved in 200 mL of water. The load provides 0.1385 mol glucose and 0.1385 mol fructose.

SUMMARY:
To investigate the secretion of gut hormones, in particular glucagon-like peptide 1 (GLP-1), after ingestion of glucose and fructose as separate monosaccharides or combined in the disaccharides sucrose and isomaltulose and the effect of acarbose in gastric bypass operated subjects and BMI-matched controls.

DETAILED DESCRIPTION:
Disaccharides such as sucrose or isomaltulose (also called palatinose) require digestion into monosaccharides (both are digested to glucose and fructose) by enzymes located in the brush border of the small intestine to be absorbed. The study will investigate the influence of carbohydrate digestion on gut hormone secretion.

ELIGIBILITY:
Gastric bypass operated patients:

Inclusion Criteria:

* uncomplicated gastric bypass surgery performed minimum 12 months prior to study

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus prior to or after gastric bypass surgery
* Pregnancy or breastfeeding
* Haemoglobin levels below 6,5 mM

Healthy control subjects:

Exclusion Criteria:

* Bariatric surgery or complicated upper abdominal surgery
* Pregnancy or breastfeeding
* Haemoglobin levels below 6,5 mM
* Co-morbidities or medicine significantly affecting glucose metabolism or appetite regulation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Within group difference in GLP-1 secretion (evaluated by iAUC). | 0-240 min following carbohydrate ingestion
  Comparison of the GLP-1 responses (evaluated by iAUC) induced by the different carbohydrate loads.

SECONDARY OUTCOMES:
Between group comparison of GLP-1 secretion (evaluated by iAUC). | 0-240 min following carbohydrate ingestion
  GLP-1 secretion (evaluated by iAUC) in gastric bypass operated patients compared to BMI-matched control subjects for each of the carbohydrate loads.
Between group comparison of differences in GLP-1 secretion (evaluated by iAUC). | 0-240 min following carbohydrate ingestion
  Differences in GLP-1 secretion (evaluated by iAUC) induced by the different carbohydrate loads in gastric bypass operated patients compared to differences in BMI-matched control subjects.
Responses (evaluated by iAUC) of glucose within and between groups. | 0-240 min following carbohydrate ingestion
Responses (evaluated by iAUC) of insulin within and between groups. | 0-240 min following carbohydrate ingestion
Responses (evaluated by iAUC) of C-Peptide within and between groups. | 0-240 min following carbohydrate ingestion
Responses (evaluated by iAUC) of peptide YY (PYY) within and between groups. | 0-240 min following carbohydrate ingestion
Responses (evaluated by iAUC) of Gastric Inhibitory Peptide (GIP) within and between groups. | 0-240 min following carbohydrate ingestion
Responses (evaluated by iAUC) of glucagon within and between groups. | 0-240 min following carbohydrate ingestion
Responses (evaluated by iAUC) of oxyntomodulin within and between groups. | 0-240 min following carbohydrate ingestion
Responses (evaluated by iAUC) of cholecystokinin (CCK) within and between groups. | 0-240 min following carbohydrate ingestion
Responses (evaluated by iAUC) of bile acids within and between groups. | 0-240 min following carbohydrate ingestion

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Endocrinology, Hvidovre, Denmark

REFERENCES:
- [Derived] Martinussen C, Bojsen-Moller KN, Dirksen C, Svane MS, Kristiansen VB, Hartmann B, Holst JJ, Madsbad S. Augmented GLP-1 Secretion as Seen After Gastric Bypass May Be Obtained by Delaying Carbohydrate Digestion. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3233-3244. doi: 10.1210/jc.2018-02661. PMID 30844053